CLINICAL TRIAL: NCT02948569
Title: Evaluation of 3-V Bioscience-2640, a FASN Inhibitor, to Reduce de Novo Lipogenesis in Subjects With Characteristics of the Metabolic Syndrome
Brief Title: Evaluation of 3-V Bioscience-2640 to Reduce de Novo Lipogenesis in Subjects With Characteristics of Metabolic Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: Sagimet Biosciences Inc. (Industry)
Responsible Party: Principal Investigator, Elizabeth Jane Parks, Professor, Nutrition & Exercise Physiology-MED, University of Missouri-Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006432
Record Dates: First submitted 2016-10-18; First posted 2016-10-28 (Estimated); Results first posted 2023-04-20 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2023-03

CONDITIONS: Metabolic Syndrome
Keywords: Obesity; Hyperlipidemia; Impaired fasting glucose; Insulin resistance; Hypertension
MeSH Terms: conditions — Metabolic Syndrome; Obesity; Hyperlipidemias; Insulin Resistance; Hypertension

STUDY DESIGN:
Masking Description: There is only one treatment arm in this study and the subjects are all aware that they are on active treatment. The outcomes assessor will be masked as to which data are from the baseline visit and which are from the follow-up visit. In other words, data will be analyzed in the lab in a blinded fashion as to whether the samples are from before or after treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 3-V Bioscience-2640 (Experimental): Subjects will take a singly daily dose of 3-V Bioscience-2640 before bedtime or 22:30, whichever comes first, for 10 days.
  Interventions: Drug: 3-V Bioscience-2640

INTERVENTIONS:
Drug: 3-V Bioscience-2640 — Subjects will take a singly daily dose of 3-V Bioscience-26400 before bedtime or 22:30, whichever comes first, for 10 days.

SUMMARY:
Metabolic syndrome increases the risk for development of heart disease. Another condition associated with metabolic syndrome is fatty liver disease which is also referred to as nonalcoholic fatty liver disease (NAFLD). Recently, drugs that block fatty acid synthesis have been developed to treat cancer. These drugs are now being considered for the treatment of NAFLD. A research test designed to measure liver fatty acid synthesis involves consumption of a sugary solution and measurement of blood fats over a six-hour period. The present study will test the drug 3-V Bioscience-2640 in healthy subjects with characteristics of the metabolic syndrome before and after 10 days of treatment to determine if 50 mg/d significantly reduces liver fat synthesis and lowers liver fat storage.

DETAILED DESCRIPTION:
The drug 3-V Bioscience-2640 has been tested previously in subjects with cancer because the lipogenesis pathway is important to the control of some cancer progression. Palmitate (C16:0), a saturated, 16-carbon fatty acid is a biomarker of lipogenesis present in blood triglyceride (TG), was found to be reduced significantly. A second biomarker of lipogenesis, malonyl carnitine, was significantly increased in patients as expected. The present study will test a lower dose (50 mg/d) than the maximum dose previously administered. Here, the subjects will be men with characteristics of the metabolic syndrome, who are otherwise healthy. The focus on subjects with metabolic syndrome is based on the fact that the future use of the drug will be in patients with NAFLD who will likely have metabolic syndrome characteristics.

In humans, the primary organ that synthesizes fatty acids is the liver, and this process occurs when simple sugars are consumed in the diet. The carbons in the sugars clear to the liver and become the molecule acetyl-Coenzyme A, which is the building block of fatty acids. The Laboratory of Elizabeth Parks, co-investigator, has developed an oral sugars tolerance test (OSTT) to determine the magnitude of liver stimulation of fatty acid synthesis when an individual consumes an oral bolus of sugars. This test involves the subject undergoing IV infusion with the stable (non-radioactive) isotope (13C1-acetate). The isotope gets incorporated into fatty acids that are being synthesized during the course of the infusion and when sugars stimulate lipogenesis, the label is more abundance. Those labeled fatty acids are detected as present in the blood very low-density lipoprotein (VLDL) component.

In the present study, the investigators will use this protocol to determine whether 10 days of drug treatment (one dose per day) will significantly reduce fasting and fructose-stimulated lipogenesis. The study is divided into 3 parts which will support the plan for minor adjustments in the dose of drug after the results from the first two research subjects are available in order to optimize the suppression of lipogenesis, while also minimizing any side effects the drug might have. The study is a repeated-measures design, with each subject serving as his own control. The study will be unblinded with respect to the research staff working directly with the subjects. However, laboratory personnel who will be running the biochemical analyses will be blinded as to whether they are analyzing baseline or post-treatment samples.

ELIGIBILITY:
Inclusion Criteria:

1. Men with characteristics of metabolic syndrome

   1. Waist circumference greater than 40 in (102 cm)
   2. Plasma TG greater than 150 mg/dL
   3. HDL cholesterol less than 40 mg/dL
   4. Blood pressure greater than or equal to 130/85 mmHg
   5. Fasting plasma glucose greater than 100 mg/dL but less than 126 mg/dL
   6. Fasting insulin great than 10 microunits/mL
2. 35-60 years of age
3. Overweight/obese subjects with BMI 27.1 - 35.0 kg/m2
4. Family history of cardiovascular disease or diabetes
5. Habitual diets containing ≥ 5.0% of energy from added sugars
6. Creatinine clearance of ≥80 mL/min

Exclusion Criteria:

1. Diagnosed cardiovascular disease (unstable angina, New York Heart Association angina > Grade 2), abnormal thyroid function or liver/kidney disease, renal dysfunction (defined by a glomerular filtration rate <80 mL/min)
2. Chronic skin disorder or treatment for acne
3. History of clinically significant dry eye or eye diseases such as glaucoma
4. Diabetes defined as fasting glucose ≥ 125 mg/dL or HbA1c ≥ 6.5%
5. Habitual diets with low content of added sugars (<5% of total energy)
6. Any tobacco use
7. Elevated liver enzymes ≥ 3x normal (regional norms Alanine transaminase <42 U/L, aspartate aminotransferase <40 U/L, and gamma-glutamyl transferase 8-61 U/L)
8. Contraindications of MRI
9. Alcohol intake weekly greater than 56 g/week (4 standard drinks/wk).
10. Major surgery or donation of blood of >500 mL within the past 8 wks.
11. Patients with uncontrolled hypertension, i.e. ≥160/95 mmHg.
12. Patients with known cardiac abnormalities.

Ages: 35 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-12-18 (Actual); Study Completion 2019-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth J Parks, PhD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Syed-Abdul MM, Parks EJ, Gaballah AH, Bingham K, Hammoud GM, Kemble G, Buckley D, McCulloch W, Manrique-Acevedo C. Fatty Acid Synthase Inhibitor TVB-2640 Reduces Hepatic de Novo Lipogenesis in Males With Metabolic Abnormalities. Hepatology. 2020 Jul;72(1):103-118. doi: 10.1002/hep.31000. Epub 2020 May 7. PMID 31630414

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment process will include the typical flyers and notices put in public spaces. All advertisements will state the purpose of the study, eligibility criteria and will tell subjects to call into our laboratory for more information. During these calls, the study will be described briefly. A checklist will be phone through to perform initial screening for age, gender, health status. Subjects who are eligible by phone screen will be scheduled for a screening visit.
Groups:
- 3-V Bioscience-2640: Subjects will take a singly daily dose of 3-V Bioscience-2640 before bedtime or 22:30, whichever comes first, for 10 days.
  3-V Bioscience-2640: Subjects will take a singly daily dose of 3-V Bioscience-2640 before bedtime or 22:30, whichever comes first, for 10 days.
Period: Overall Study
Arm/Group | 3-V Bioscience-2640
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 3-V Bioscience-2640
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.1 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in Hepatic Lipogenesis
Description: Subject undergoes a stable isotope infusion followed by blood draws. Plasma lipid samples are measured by gas chromatography/mass spectrophotometry.
Time Frame: Baseline and after 10 days of treatment
Measure: Mean (Standard Error); unit: abs percent change fasting lipogenesis
Arm/Group | 3-V Bioscience-2640
Number analyzed (Participants) | 12
abs percent change fasting lipogenesis | 5.6 (1.5)

2. Secondary Outcome: Change in Liver Fat Measured by MRI
Description: Subject undergoes MRI of abdomen to quantify liver fat.
Time Frame: Baseline and 10 days of treatment
Measure: Mean (Standard Error); unit: absolute percent change in liver fat
Arm/Group | 3-V Bioscience-2640
Number analyzed (Participants) | 12
absolute percent change in liver fat | 1.8 (1.2)

3. Secondary Outcome: Change in Skin Sebum Production
Description: Subjects will undergo a skin test in which 4 pieces of clear Sebutape will be placed on the forehead for 30 minutes. The tape is then removed with a sample of sebum (skin oils). The tape is shipped to a lab for processing where lipid content will be analyzed.
Time Frame: Baseline and 10 days of treatment
Measure: Mean (Standard Error); unit: Absolute change sebum TG (nmol/sample))
Arm/Group | 3-V Bioscience-2640
Number analyzed (Participants) | 6
Absolute change sebum TG (nmol/sample)) | 6.76 (2.08)

ADVERSE EVENTS:
Time Frame: 20 days
Description: The following adverse events were queried at screening and during the 6 study visits over 20 days.
  1. Disturbed bowel habits
  2. Constipation
  3. Diarrhea
  4. Dry mouth
  5. Dry skin
  6. Fatigue
  7. Flatulence
  8. Hair loss
  9. Headache
  10. Itching
  11. Loss of appetite
  12. Nausea and vomiting
  13. Sleep disturbances
  14. Tiredness
Arm/Group | 3-V Bioscience-2640
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 2/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3-V Bioscience-2640 (N=12)
hair loss (Skin and subcutaneous tissue disorders) | 2 (2) — The possibility of hair loss is listed in the consent form and, given that the effect of this drug is to lower body oil synthesis, the mechanism for this AE is likely a reduction in the oil production at the base of the hair follicle.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-03-08): https://cdn.clinicaltrials.gov/large-docs/69/NCT02948569/Prot_SAP_ICF_002.pdf